CLINICAL TRIAL: NCT01895166
Title: Diagnostic Value of Endobronchial Ultrasound(EBUS) With a Guide Sheath(GS) for Peripheral Pulmonary Lesions(PPLs) Without Fluoroscopy: a Randomized Controlled Trial
Brief Title: EBUS-GS-TBLB With or Without Fluoroscopy for the Diagnosis of PPLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Fukushima Medical University (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Endoscope Center, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201301
Record Dates: First submitted 2013-03-25; First posted 2013-07-10 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer
Keywords: Endobronchial ultrasonography with a guide sheath; Peripheral pulmonary lesions; Transbronchial biopsy
MeSH Terms: conditions — Lung Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBUS-GS group (Experimental): The EBUS probe and GS are confirmed to reach the lesion by EBUS images alone, cytologic and pathologic specimens are obtained without fluoroscopic guidance.
  Interventions: Procedure: EBUS-GS
- EBUS-GS-X-ray group (Active Comparator): The EBUS probe and GS are confirmed to reach the lesion by EBUS images and radiograph fluoroscopy, cytologic and pathologic specimens are obtained under fluoroscopic guidance.
  Interventions: Procedure: EBUS-GS; Procedure: X-ray

INTERVENTIONS:
Procedure: EBUS-GS — EBUS is performed using an endoscope ultrasound system , which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm and a GS (K-201; Olympus).
Procedure: X-ray — The radiograph fluoroscopy are performed when the probe and GS are confirmed to reach the lesion by EBUS images ,cytologic and pathologic specimens are obtained under fluoroscopic guidance.
  Arms: EBUS-GS-X-ray group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of endobronchial ultrasound-guide sheath(EBUS-GS) for the diagnosis of peripheral pulmonary lesions (PPLs) without radiographic fluoroscopy.

DETAILED DESCRIPTION:
The investigators evaluated the efficacy and safety of transbronchial biopsy (TBB) and bronchial brushing by endobronchial ultrasonography (EBUS) with a guide sheath (GS) as a guide for diagnosing peripheral pulmonary lesions (PPLs) without radiographic fluoroscopy.The study is designed as a two-center prospective randomized controlled trial. The participating centers are Department of pulmonary medicine and endoscope center, Shanghai chest Hospital affiliated to Shanghai JiaoTong University School, China. Department of pulmonary medicine, Fukushima Medical University, Japan.Patients are divided into two groups, EBUS-GS-X-ray group and EBUS-GS group.Each subject will be randomized to each group.The study is expected to enroll 100 patients at 2 centers (China:75, Fukushima:25).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals eligible for inclusion are patients that the CT scan appearance of the PPLs showed the longest diameter was more than 2 cm and solid lesions.

Exclusion Criteria:

1. The lesion is close to the pleural membrane
2. Refusal of participation
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The difference of diagnostic value of EBUS-GS-TBLB with fluoroscopy as compared to EBUS-GS-TBLB alone | Up to half year
  The diagnostic value mean sensitivity and specificity in two groups

SECONDARY OUTCOMES:
The difference of complications of EBUS-GS-TBLB with fluoroscopy as compared to EBUS-GS-TBLB alone | Up to half year
  Complications mean a composite of operation-related serious adverse events (pneumothorax, bleeding, etc.) during and after the operation in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

REFERENCES:
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Background] Yoshikawa M, Sukoh N, Yamazaki K, Kanazawa K, Fukumoto S, Harada M, Kikuchi E, Munakata M, Nishimura M, Isobe H. Diagnostic value of endobronchial ultrasonography with a guide sheath for peripheral pulmonary lesions without X-ray fluoroscopy. Chest. 2007 Jun;131(6):1788-93. doi: 10.1378/chest.06-2506. PMID 17565021
- [Background] Yamada N, Yamazaki K, Kurimoto N, Asahina H, Kikuchi E, Shinagawa N, Oizumi S, Nishimura M. Factors related to diagnostic yield of transbronchial biopsy using endobronchial ultrasonography with a guide sheath in small peripheral pulmonary lesions. Chest. 2007 Aug;132(2):603-8. doi: 10.1378/chest.07-0637. Epub 2007 Jun 15. PMID 17573504
- [Background] Steinfort DP, Khor YH, Manser RL, Irving LB. Radial probe endobronchial ultrasound for the diagnosis of peripheral lung cancer: systematic review and meta-analysis. Eur Respir J. 2011 Apr;37(4):902-10. doi: 10.1183/09031936.00075310. Epub 2010 Aug 6. PMID 20693253